CLINICAL TRIAL: NCT02630719
Title: Timolol Eye Drops in the Treatment of Acute Migraine Headache
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll sufficient participants
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: Truman Medical Center (Other)
Responsible Party: Principal Investigator, Sean Gratton, Assistant Professor and Staff Physician, University of Missouri, Kansas City
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 15-152; #15-060 (Other: Truman Medical Center)
Record Dates: First submitted 2015-11-25; First posted 2015-12-15 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Migraine
Keywords: headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Timolol eye drops (Active Comparator): All subjects received timolol eye drops or placebo (artificial tears) for two months then crossed over to the opposite medication for the final two months of the study.
  Interventions: Drug: Timolol eye drops
- Artificial tears (Placebo Comparator): All subjects received timolol eye drops or placebo (artificial tears) for two months then crossed over to the opposite medication for the final two months of the study.
  Interventions: Drug: Artificial tears

INTERVENTIONS:
Drug: Timolol eye drops — eye drops
  Arms: Timolol eye drops
Drug: Artificial tears — Placebo drop
  Arms: Artificial tears

SUMMARY:
The goal of this study is to determine whether timolol eye drops are effective in alleviating acute migraine headaches. Subjects will be randomized to receive either timolol eye drops or placebo (tears) to use as a migraine abortive medication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine headache

Exclusion Criteria

* Non-migraine headache
* Use of systemic beta-blocker
* Medical history of hypotension, bradycardia, syncope or other significant cardiovascular disease
* Medical history of difficulty breathing, asthma or chronic obstructive pulmonary disease or other pulmonary disease
* Medical history of glaucoma, ocular hypertension or hypotony, punctual stenosis, current use of other ophthalmic medications
* Previous adverse reaction to timolol or other beta-blockers
* Inability to self-administer eye drop due to physical or cognitive disorders
* Currently pregnant or breastfeeding
* Pregnant in the past year
* Non-english speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Gratton, MD, Principal Investigator — UMKC
Locations (1):
- Truman Medical Center, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Cossack M, Nabrinsky E, Turner H, Abraham A, Gratton S. Timolol Eyedrops in the Treatment of Acute Migraine Attacks: A Randomized Crossover Study. JAMA Neurol. 2018 Aug 1;75(8):1024-1025. doi: 10.1001/jamaneurol.2018.0970. PMID 29799915

RESULTS

PARTICIPANT FLOW:
Groups:
- Timolol Eye Drops First: Timolol ophthalmic solution 0.5% first, then Artificial Tears
  Subjects instill one drop of the solution at the onset of headache into both eyes. Subjects may repeat with one more drop into each eye after 30 minutes.
  Each intervention period is 2 months with a 4 day washout period in between.
- Artificial Tears First: Artificial tears first, then timolol ophthalmic solution 0.5%
  Subjects instill one drop of the solution at the onset of headache into both eyes. Subjects may repeat with one more drop into each eye after 30 minutes.
  Each intervention period is 2 months with a 4 day washout period in between.
Period: Overall Study
Arm/Group | Timolol Eye Drops First | Artificial Tears First
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Timolol Eye Drops First: Treatment with timolol eye drops at the onset of an acute migraine headache for the first 2 months, then a 4 day washout period, followed by Artificial tears at the onset of an acute migraine headache for the next 2 months.
  Subjects instill one drop of the solution at the onset of headache into both eyes. Subjects may repeat with one more drop into each eye after 30 minutes.
- Artifical Tears First: Treatment with artificial eye drops at the onset of an acute migraine headache for the first 2 months, then a 4 day washout period, followed by timolol eye drops at the onset of an acute migraine headache for the next 2 months.
  Subjects instill one drop of the solution at the onset of headache into both eyes. Subjects may repeat with one more drop into each eye after 30 minutes.
- Total: Total of all reporting groups
Arm/Group | Timolol Eye Drops First | Artifical Tears First | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 6 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Timolol Eye Drops in the Treatment of Acute Migraine Headache
Description: Percent of migraine attacks at 0 or 1 on the 4-point Rating Scale recommended by the International Headache Society:
  0: no headache
  1. mild headache
  2. moderate headaches
  3. severe headache
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage of migraine attacks at 0 or 1
Groups:
- Timolol Eye Drops: Treatment with timolol eye drops at the onset of an acute migraine headache
  Timolol eye drops: eye drops
- Artificial Tears: Treatment with artificial eye drops at the onset of an acute migraine headache
  Artificial tears: Placebo drop
Arm/Group | Timolol Eye Drops | Artificial Tears
Number analyzed (Participants) | 10 | 10
percentage of migraine attacks at 0 or 1 | 78 (31) | 67 (30)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Timolol Eye Drops | Artificial Tears
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Informed Consent Form (2016-08-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT02630719/ICF_000.pdf
  • Study Protocol (2015-03-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT02630719/Prot_001.pdf
  • Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT02630719/SAP_002.pdf